CLINICAL TRIAL: NCT06336824
Title: Early Intravenous to Oral Antibiotic Switch in Uncomplicated Staphylococcus Aureus Bacteraemia: The EVOS Randomized Controlled Trial
Brief Title: Early Intravenous to Oral Antibiotic Switch in Uncomplicated Staphylococcus Aureus Bacteraemia
Acronym: EVOS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Clinical Research Centre, Malaysia (Other)
Responsible Party: Principal Investigator, Steven Lim Chee Loon, Infectious Diseases Physician, Ministry of Health, Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EVOS 1.3 dated 12 March 2024
Record Dates: First submitted 2024-03-22; First posted 2024-03-29 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Staphylococcus Aureus Bacteremia
Keywords: bacteremia; oral antibiotics; Staphylococcus aureus
MeSH Terms: conditions — Bacteremia; Staphylococcal Infections | interventions — Trimethoprim, Sulfamethoxazole Drug Combination; Clindamycin; Linezolid; Cloxacillin; Cefazolin; Vancomycin; Ceftaroline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early Oral Switch Therapy (EOS) (Experimental): Patients will switch from IV therapy to oral antibiotics for 7 to 11 days to achieve a total 14 days of definitive antimicrobial therapy for SAB.
  First choice oral antibiotics for MSSA and MRSA: Tab. Trimethoprim-sulfamethoxazole (TMP 10mg/kg/day)
  Alternative oral antibiotics for MSSA: Tab. Clindamycin 600mg TDS, Tab. Cephalexin 1gm QID, Tab Linezolid 600mg BD
  Alternative oral antibiotics for MRSA: Tab. Linezolid 600mg BD
  Interventions: Drug: Tab. Trimethoprim-sulfamethoxazole, Tab. Clindamycin, Tab. Cephalexin, or Tab. Linezolid
- Standard IV therapy (SIV) (Active Comparator): Patients will continue with IV therapy for 7 to 11 days to achieve a total 14 days of definitive antimicrobial therapy for SAB.
  First choice IV antibiotics for MSSA: IV Cloxacillin 2g every 4 or 6 hours
  Alternative IV antibiotics for MSSA: IV Cefazolin 2g TDS
  First choice IV antibiotics for MRSA: IV Vancomycin 15-20mg/kg BD
  Alternative IV antibiotics for MRSA: IV Ceftaroline 600mg TDS
  Interventions: Drug: IV Cloxacillin, IV Cefazolin, IV Vancomycin, or IV Ceftaroline

INTERVENTIONS:
Drug: Tab. Trimethoprim-sulfamethoxazole, Tab. Clindamycin, Tab. Cephalexin, or Tab. Linezolid — The choice of study drug will depend on the susceptibility of the respective isolate, expected drug interactions, contraindications, and expected side effects.
  Investigators will assess whether the "first-choice" regimen can be given and then consider the alternative regimen. The antibiotics can be switched from first choice to the respective alternative medications during the intervention period if clinically necessary. The route of administration must be maintained according to the randomized group.
  Other Names: Bactrim; Dalacin; Ospexin; Zyvox
  Arms: Early Oral Switch Therapy (EOS)
Drug: IV Cloxacillin, IV Cefazolin, IV Vancomycin, or IV Ceftaroline — The choice of study drug will depend on the susceptibility of the respective isolate, expected drug interactions, contraindications, and expected side effects.
  Investigators will assess whether the "first-choice" regimen can be given and then consider the alternative regimen. The antibiotics can be switched from first choice to the respective alternative medications during the intervention period if clinically necessary. The route of administration must be maintained according to the randomized group.
  Other Names: Cloxacillin Sodium; Cefazolin Sandoz; Vancotex; Zinforo
  Arms: Standard IV therapy (SIV)

SUMMARY:
The Early Intravenous to Oral Antibiotic Switch in Uncomplicated Staphylococcus aureus Bacteraemia (EVOS) study is a multicentre, randomized, open-label, parallel group, phase 3, non-inferiority trial of early intravenous to oral antibiotic switch in comparison with standard intravenous antibiotic regime among patients with uncomplicated Staphylococcus aureus bacteraemia (SAB). The study is based on the hypothesis that an early switch from IV to oral antimicrobial therapy is non-inferior and safe compared to conventional minimum 14-day course of IV therapy in patients with low-risk uncomplicated SAB.

DETAILED DESCRIPTION:
The study is conducted at 12 government tertiary hospitals with infectious diseases physicians in Malaysia. The study population comprises of 290 patients with uncomplicated SAB who have received 3 to 7 days of definitive IV antimicrobial therapy. Eligible participants are randomized 1:1 into 2 groups, early oral antibiotic switch versus standard IV antibiotic therapy, following the inclusion and exclusion criteria.

The study consists of 3 stages for each patient with a duration of approximately 12 weeks: screening and enrolment, open-label treatment with 7 to 11 days of study antibiotics, and follow-up until day 90 post-randomization. Phone call or inpatient follow up will be conducted at Day 7-11, Day 30, and Day 90 post- randomization to review patient's condition.

ELIGIBILITY:
Inclusion Criteria:

1. Blood culture positive for Staphylococcus aureus (S. aureus).
2. Received 3 to 7 days of definitive IV antimicrobial therapy, defined as:

   * Cloxacillin or cefazolin for methicillin-sensitive staphylococcus aureus (MSSA); Vancomycin or ceftaroline for methicillin-resistant staphylococcus aureus (MRSA).
   * Proven in-vitro susceptibility and adequate dosing given (as determined by the principal investigator).
3. Achieved clearance of bacteraemia, defined as at least one documented latest negative follow-up blood culture obtained within 72 hours after the initiation of definitive IV antimicrobial therapy.
4. Achieved defervescence, defined as sustained body temperature ≤37.5°C within 48 hours before randomization.
5. Able to provide written informed consent to participate trial.

Exclusion Criteria:

1. Evidence of metastatic infection of S. aureus: for example, infective endocarditis, intraabdominal abscess, lung empyema, and osteomyelitis. Radiological investigations such as chest X-ray, ultrasound, echocardiogram, and CT scan are not mandatory prior to enrolment, but should be done at the discretion of the treating physician if clinically indicated.
2. Septic shock, defined as hypotension requiring vasopressors to maintain MAP ≥65 mmHg despite adequate volume resuscitation.
3. Received more than 5 days of non-study antibiotics as empirical therapy prior to enrolment.
4. Polymicrobial bloodstream infection, defined as isolation of pathogens other than S. aureus from a blood culture obtained prior to randomization. Common skin contaminants such as coagulase-negative staphylococci, Bacillus spp., and diphtheroid will not be considered to represent polymicrobial infection.
5. Known history of S. aureus infection within the past 3 months.
6. Inability to tolerate oral therapy or poor absorption of oral medications, or not suitable for ongoing IV therapy (for example, difficult intravenous access)
7. No options of oral antibiotic available for patient due to:

   * In vitro resistance of S. aureus to all oral study drugs.
   * Known contraindications to receive the active oral study drugs. For example, hypersensitivity reaction to trimethoprim-sulfamethoxazole, thrombocytopenia secondary to linezolid etc.
   * Non-availability of oral study drugs at the study sites.
8. Patient is concomitantly receiving oral antibiotics which are active against S. aureus. For example, trimethoprim-sulfamethoxazole for Pneumocystis jirovecii pneumonia prophylaxis.
9. Presence of a non-removable foreign body such as prosthetic heart valve, vascular graft, pacemaker, automated implantable cardioverter-defibrillator, ventriculoperitoneal shunt, prosthetic joint, and fracture fixation implant
10. Failure or inability to remove intravascular catheter that is present when first positive blood culture was drawn.
11. Known comorbidity that increased the risk of complicated infections:

    * End-stage renal disease
    * Severe liver disease (Child-Pugh class C)
    * Severe immunodeficiency:

      * HIV-positive patients with CD4<200 cells/uL or AIDS
      * primary immunodeficiency disorders
      * high-dose steroid therapy (>1 mg/kg prednisone or equivalent doses given for > 4 weeks or planned during intervention)
      * immunosuppressive therapy
      * neutropenia (<500 neutrophils/μl) at randomization or neutropenia expected during intervention phase due to immunosuppressive treatment
      * solid organ or hematopoietic stem cell transplantation within the past 6 months or planned during treatment period

13.Short life expectancy < 3 months

14.Pregnancy (for women of childbearing potential)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2024-06-28 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Rate of SAB-relapse | 90 days
  defined as any new positive blood culture with S. aureus, and/or newly diagnosed metastatic S. aureus infection resulting from hematogenous dissemination

SECONDARY OUTCOMES:
Number of days of hospitalization | 90 days
  Number of calendar days of hospitalisation after the first positive blood culture for S. aureus.
Rate of all-cause mortality | 90 days
  Any death occurred within 90 days of randomization.
Rate of complications related to IV therapy | 90 days
  Any complications related to insertion or usage of peripheral branula or central catheter, and administration of IV drugs
Rate of Clostridium difficile diarrhoea | 90 days
  A diagnosis of diarrhoea with ≥1 stool sample tested positive for C. difficile toxin or toxin gene.
Rate of adverse events | 30 days
  Any untoward medical occurrence in a subject administered a medicinal product and which does not necessarily have a causal relationship with treatment.

CONTACTS AND LOCATIONS:
Locations (12):
- Malaysia (12):
  - Hospital Sultanah Aminah, Johor Bahru, Johor
  - Hospital Sultanah Bahiyah, Alor Star, Kedah
  - Hospital Sultan Abdul Halim, Sungai Petani, Kedah
  - Hospital Tuanku Ja'afar, Seremban, Negeri Sembilan
  - Hospital Raja Permaisuri Bainun, Ipoh, Perak
  - Hospital Pulau Pinang, George Town, Pulau Pinang
  - Hospital Seberang Jaya, Seberang Jaya, Pulau Pinang
  - Hospital Ampang, Ampang, Selangor
  - Hospital Sultan Idris Shah Serdang, Kajang, Selangor
  - Hospital Tengku Ampuan Rahimah, Klang, Selangor
  - Hospital Selayang, Selayang Baru Utara, Selangor
  - Hospital Melaka, Malacca

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-12): https://cdn.clinicaltrials.gov/large-docs/24/NCT06336824/Prot_SAP_002.pdf